CLINICAL TRIAL: NCT02978612
Title: Adjuvant Chemotherapy In Elderly With Colon Cancer Stage III - Geriatric Assessment and Prognostic Gene Signatures
Brief Title: Adjuvant Chemotherapy In Elderly With Colon Cancer Stage III
Acronym: ACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Marianne Grønlie Guren, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1252
Record Dates: First submitted 2016-06-15; First posted 2016-12-01 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Colon Cancer
Keywords: Colorectal Neoplasms
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm Capecitabine (Experimental): Capecitabine 1000 mg/m2 bid day 1-14 q3 weeks, 8 cycles
  Interventions: Drug: Capecitabine
- Arm No treatment (No Intervention): no chemotherapy, observation

INTERVENTIONS:
Drug: Capecitabine — Capecitabine is a prodrug to 5-fluorouracil. It is used for adjuvant chemotherapy after surgery for colon cancer. The tablets are either 150 mg or 500 mg
  Other Names: Xeloda
  Arms: Arm Capecitabine

SUMMARY:
This is a phase 2, randomized study where the aim of the study is to investigate the tolerance of adjuvant chemotherapy, measured by functional decline, after surgery for colon cancer stage III in elderly patients. Secondary aims are disease-free survival, toxicity, late functional outcome, quality of life, to establish a geriatric assessment for selection of patients, and to examine the prognostic value of gene signature tests / biomarkers for stage III colon cancer.

DETAILED DESCRIPTION:
Patients ≥ 75 years who have undergone surgery for colon cancer stage III, are eligible for inclusion in the study. Non-eligibility includes patients with obvious impaired cognitive or physical function or patients living in nursing homes. After signing informed consent, the patients first undergo geriatric assessment. Patients that are classified as having fit or intermediate function, and with no significant cardiovascular disease, are randomized with a 2:1 randomization process to either chemotherapy (Arm A: Capecitabine 1000 mg/m2 bid day 1-14 q3 weeks, 8 cycles) or no chemotherapy (Arm B: observation).

The purpose of this study is to examine the tolerability of chemotherapy in elderly (> 75 years) patients operated on for colon cancer stage III. There is little evidence of benefit and tolerability of this therapy in the elderly; it is recommended individual consideration in elderly. In the study, a comprehensive geriatric a comprehensive geriatric assessment is performed first, to exclude frail patients or patients with serious comorbidities such as cardiovascular disease. Fit or intermediate patients will then be randomized so that 2/3 will receive chemotherapy with capecitabine tablets for 6 months, and 1/3 will not receive chemotherapy. A new geriatric assessment is performed after 6 and 12 months. The main objective of the study is to examine whether chemotherapy leads to significant loss of function, but secondary aims include survival, quality of life, and prognostic effect of biomarkers. The study may provide useful information on selection of patients who tolerate and benefit from adjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Radical surgery (R0/R1) for colon cancer
* Histologically verified adenocarcinoma of the colon
* Histologically verified lymph node metastases (Stage III)
* Age ≥ 75 years
* Able to undergo ambulatory treatment (adequate physical and mental function)
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to The International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH GCP) and national regulations.

Exclusion Criteria:

* Distant metastases (stage IV)
* Frail according to geriatric assessment
* Significant cardiovascular disease (congestive heart failure, symptomatic coronary artery disease and cardiac dysrhythmia) or myocardial infarction within the past 12 months
* Previous treatment with chemotherapy for colorectal cancer
* Metastatic disease from other cancer
* Reduced cognitive function not enabling ability to give informed consent or compliance with the study
* History of prior or concurrent malignant neoplasm other than colorectal adenocarcinoma within the past five years, except curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix
* Adverse reactions or hypersensitivity to capecitabine or related drugs and/or its excipients. Need to use medications contraindicated according to SmPC of the IMP(s), such as sorivudine, brivudin or chemically related compounds. Any other contraindication listed on the summary of product characteristics (SmPC) of the investigational medicinal Product (IMP)
* Use of methotrexate or other cytotoxic drugs as treatment of rheumatoid arthritis or other inflammatory disease and where it is considered contraindicated to stop this medication
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Any reason why, in the opinion of the investigator, the patient should not participate

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
Functional decline in instrumental activities of daily living (IADL) and/or activities of daily living (ADL) | 1 year after surgery
  Tolerance of adjuvant chemotherapy in elderly patients, measured as functional decline or independency, by ADL and IADL questionnaires.

SECONDARY OUTCOMES:
Relative dose intensity; i.e the percentage of planned chemotherapy dose the patient actually receives | through study completion
  Number of planned chemotherapy cycles given, total dose given
Toxicity of chemotherapy | During treatment and follow-up 1 year after surgery
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Disease-free survival | 3 years after surgery
  Follow-up, 3-year disease-free survival
Quality of life questionnaire 1 | Time of randomization, 6 months and 1 year after surgery
  EQ-5D-5L
Quality of life questionnaire 2 | Time of randomization, 6 months and 1 year after surgery
  EORTC QLQ-C30
Quality of life questionnaire 3 | Time of randomization, 6 months and 1 year after surgery
  QLQ-ELD14
Validation of the performance of prognostic biomarkers in estimating disease-free survival | 3 years after surgery
  Prognostic biomarkers validated for performance in estimating 3-year disease-free survival
Overall survival | 5 years after surgery
  Follow-up, 5-year disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Marianne G Guren, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided